CLINICAL TRIAL: NCT05456100
Title: A Randomized Controlled Trial Testing Expressive Helping for Chinese American Cancer Survivors
Brief Title: Chinese American Cancer Survivors Writing Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20-0603; 1K01MD014750 (NIH)
Record Dates: First submitted 2022-07-06; First posted 2022-07-13 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Expressive Helping (Experimental): Participants complete a 20-minute expressive writing session once per week for the first three weeks. During Week 4, participants complete a 20-minute peer support writing session.
  Interventions: Behavioral: Expressive Helping
- Expressive Writing (Active Comparator): Participants complete a 20-minute expressive writing session once per week for four weeks.
  Interventions: Behavioral: Expressive Writing
- Factual Writing (Active Comparator): Participants complete a 20-minute factual writing about their cancer diagnosis and treatment every week for four weeks.
  Interventions: Behavioral: Factual Writing

INTERVENTIONS:
Behavioral: Expressive Helping — Expressive helping involves a combination of emotional disclosure and peer support writing completed over four weeks.
  Arms: Expressive Helping
Behavioral: Expressive Writing — Expressive writing involves emotional disclosure writing over four weeks.
  Arms: Expressive Writing
Behavioral: Factual Writing — Factual writing involves writing facts about cancer treatment and experiences over four weeks.
  Arms: Factual Writing

SUMMARY:
The Chinese American Cancer Survivors Writing Study is a Randomized Controlled Trial (RCT) testing the feasibility and efficacy of the Expressive Helping (EH) intervention among Chinese American cancer survivors.

DETAILED DESCRIPTION:
Chinese Americans are one of the fastest growing immigrant groups in the United States, but there is still a lack of culturally-sensitive and linguistically-appropriate resources and interventions for this group. To address this gap, the investigators will examine the efficacy and feasibility of Expressive Helping, a writing intervention designed to lead participants to write about their cancer experiences. Participants will be adult cancer survivors of Chinese descent. After screening and consent, eligible participants will be enrolled in a 1:1:1 randomized controlled trial. Assessments of psychological symptoms will occur at baseline (prior to randomization), 1-month post-intervention, 3-months post-intervention, and 6-months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old.
* Prefer speaking in Mandarin Chinese or Cantonese, and able to read and write Simplified or Traditional Chinese.
* Within 5 years after completing primary treatment or have completed primary treatment but still on medication for managing cancer-related symptoms.

Exclusion Criteria:

* Difficulties with writing
* Current active participation in support groups (i.e., attending more than once per week)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-07-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rates | through study completion, an average of 6 months
  The number of participants screened for eligibility, percent eligible to participate, and percent of people who refuse to participate will be tracked.
Retention rates | through study completion, an average of 6 months
  Percent of participants who complete each stage of the study (e.g., baseline survey, writing sessions, follow-ups) will be tracked.
Completion rate of writing sessions | through study completion, an average of 6 months
  Assessed by dividing the number of writing sessions finished by the number of sessions assigned.

SECONDARY OUTCOMES:
Changes in depressive symptoms assessed by the Center for Epidemiologic Studies Depression Scale | Baseline to 1-month follow-up, 3-month follow-up, and 6-month follow-up
  Depressive symptoms will be measured with the 10-item Center for Epidemiologic Studies Depression Scale (CES-D). The score can range from 0-30 and higher scores indicate more depressive symptoms.
Changes in anxiety symptoms assessed by the Generalized Anxiety Disorder Screener | Baseline to 1-month follow-up, 3-month follow-up, and 6-month follow-up
  Anxiety symptoms will be measured with the 7-item GAD-7 scale (Spitzer et al., 2006). This scale measures generalized anxiety symptoms in the past 7 days, has score ranges from 0-21 with higher scores indicating greater anxiety symptoms.
Changes in health-related quality of life assessed by the Functional Assessment of Cancer Therapy: General (FACT-G). | Baseline to 1-month follow-up, 3-month follow-up, and 6-month follow-up
  Health-related quality of life will be measured by the 27-item FACT-G, which assess four domains: physical well-being, social well-being, emotional well-being and functional well-being. The score ranges from 0-108 with higher scores indicating better quality of life.
Changes in perceived stress assessed by the Perceived Stress Scale. | Baseline to 1-month follow-up, 3-month follow-up, and 6-month follow-up
  Perceived stress is measured by the 10-item Perceived Stress Scale (PSS). The score ranges from 0-40 with higher scores indicating higher perceived stress.
Changes in cancer-related fatigue assessed by the Functional Assessment of Chronic Illness Therapy - Fatigue | Baseline to 1-month follow-up, 3-month follow-up, and 6-month follow-up
  Cancer-related fatigue is measured by the 13-item Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT). The score ranges from 0-52 with higher scores indicating greater fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- New York University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
All IPD will be protected and maintained by the study team

DOCUMENTS (1):
  • Informed Consent Form (2025-01-24): https://cdn.clinicaltrials.gov/large-docs/00/NCT05456100/ICF_000.pdf